CLINICAL TRIAL: NCT06721091
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study Investigating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Doses of VNA-318 in Healthy Male Subjects
Brief Title: Safety, Tolerability, and Dose Response of VNA-318 in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VANDRIA (Industry)
Collaborators: Biotrial (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: VNA-318-01
Record Dates: First submitted 2024-11-20; First posted 2024-12-06 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1 (SAD): Active (Experimental): Single oral dose of VNA-318
  Interventions: Drug: VNA-318
- Part 1 (SAD): Placebo (Placebo Comparator): Single oral dose of Matching Placebo
  Interventions: Drug: Placebo
- Part 2 (MAD): Active (Experimental): Multiple oral doses of VNA-318
  Interventions: Drug: VNA-318
- Part 2 (MAD): Placebo (Placebo Comparator): Multiple oral doses of Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VNA-318 — Part 1 will consist of administration of VNA-318 at the doses of 5 mg to 180 mg in 5 to 8 successive cohorts.
  Part 2 will consist of administration of VNA-318 in 3 to 4 successive cohorts. The doses will be selected based on safety and tolerability assessments, as well as PK and, if applicable, PD data from SAD.
  Once PK suggests that the therapeutic dose has been reached in the SAD part, the SAD and MAD parts of the study could be run in parallel.
  Arms: Part 1 (SAD): Active; Part 2 (MAD): Active
Drug: Placebo — Part 1 (SAD) will consist of administration of matching placebo at the doses of 5 mg to 180 mg in 5 to 8 successive cohorts.
  Part 2 (MAD) will consist of administration of matching placebo in 3 to 4 successive cohorts. The doses will be selected based on safety and tolerability assessments, as well as PK and, if applicable, PD data from SAD.
  Arms: Part 1 (SAD): Placebo; Part 2 (MAD): Placebo

SUMMARY:
This is a phase 1, randomized, double-blind, placebo-controlled study investigating the safety, tolerability, pharmacokinetics, and pharmacodynamics of single ascending doses (SAD) and multiple ascending doses (MAD) of VNA-318 in healthy male subjects.

DETAILED DESCRIPTION:
The First-in-Human phase I, single center study investigating VNA-318, administered orally, will consist of 2 parts:

* Part 1 SAD, conducted in 5 to 8 cohorts of 8 healthy male subjects per dose level, including one optional exploratory cohort with cerebrospinal fluid (CSF) sampling
* Part 2 MAD, conducted in 3 to 4 cohorts of 12 healthy male subjects per dose level Subjects will be included in either Part 1 or 2.

A Study Safety Committee is involved and will make recommendations on the study advancement, i.e. the dose for the next planned cohort.

The doses of the MAD part will be selected by this Study Safety Committee and will be based upon safety and tolerability assessments, the observed PK and, if available and applicable, PD data from SAD.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects able and willing to provide written informed consent prior any other clinical study procedures.
2. Subjects able and willing to comply with the clinical study protocol (hospitalization periods, scheduled visits, IMP administration, clinical laboratory tests, and other study procedures including lifestyle considerations) according to International Council of Harmonization (ICH) and local regulations.

   Demography
3. Healthy male.
4. Aged 18-65 years (inclusive) on the day of signing the informed consent form (ICF). - Aged 18-45 years (inclusive) for the SAD optional exploratory cohort with CSF sampling
5. Have a body mass index (BMI) between 18.5-30.0 kg/m2 (inclusive) at screening and D 1.

   Health Status
6. Have normal physical examination and vital signs (VS) results within normal ranges at screening and D˗1. If outside normal ranges, it must be considered by the Investigator without clinically significant abnormal findings.
7. Have a clinical laboratory of blood and urine within normal ranges at screening and D-1. If outside normal ranges, it must be considered by the Investigator without clinically significant abnormal findings.
8. Have 12-lead ECG results without clinically significant abnormal findings confirmed by the Investigator at screening and D-1.
9. Non-smoker (and no other nicotine use) as determined by history (no nicotine use over the past 6 months) and by urine cotinine concentration (< 200 ng/mL) at screening and D-1.

   Contraception
10. If sexually active and not sterile, with a woman of childbearing potential, the subject and his partner must commit to using a highly effective method of birth control starting at screening and throughout the entire study and for 90 days after last dose of IMP administration:

    * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, started at least 4 weeks prior to the dosing (D1) and use of condom for the male partner.
    * Progestogen-only hormonal contraception associated with inhibition of ovulation, started at least 4 weeks prior to the dosing (D1) and use of condom for the male partner.
    * Intrauterine device placed at least 4 weeks prior to the dosing (D1), and use of condom for the male partner.
    * Intrauterine hormone-releasing system placed at least 4 weeks prior to the dosing (D1), and use of condom for the male partner.
    * Simultaneous use of a diaphragm or cervical cap with intravaginally applied spermicide and, for the male partner, a male condom.
    * Sexual abstinence (when in line with the preferred and usual subject's lifestyle).
    * Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) is not acceptable.

    Or subject with a male partner.
11. Male subjects must agree to abstain from sperm donation starting at screening and throughout the study and for 90 days following their last dose of IMP administration.

    Regulations
12. Covered by a health insurance system where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research.
13. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted.

Exclusion Criteria:

Medical History

1. Any condition or disease detected during the medical interview/physical examination that could relapse during or immediately after the study, or would render the subject unsuitable for the study, place the subject at undue risk, or interfere with the ability of the subject to complete the clinical study, as determined by the Investigator.
2. Have a history of and/or current clinically significant disease/disorder determined by the Investigator: gastrointestinal, endocrine, renal, hepatic, immunological, cardiovascular, hematological, respiratory, neurologic, metabolic, urologic, dermatologic, psychiatric disorder, or allergic disease, hypersensitivity, or allergic reactions excluding mild asymptomatic seasonal allergies (either spontaneous or following drug administration), or malignancy (including lymphoma, leukemia, and skin cancer) unless remission over 10 years.
3. Have a personal or family history of prolonged QT interval syndrome or Torsade de Pointes, or family history of sudden death.
4. Have current presence of an illness, such as a common cold, isolated headache, diarrhea, etc., within 14 days prior to D1 that is categorized as clinically significant by the Investigator.
5. History or presence of regular use of recreational or illicit drugs within 1 year before study D1.
6. Donation of blood or blood loss (i.e., > 450 ml) within 90 days, or donated plasma within 7 days prior to D-1.
7. Known significant hypersensitivity or other contraindication to any of the components of the study drug.
8. History of suicidal behavior or any risk of suicidal behavior in the opinion of a certified clinician or as evidenced by a "yes" to any questions of Columbia-Suicide Severity Rating Scale (C-SSRS) taken at screening (MAD part only).
9. Confirmed coronavirus disease 2019 (COVID-19) infection within 90 days of screening or contact with an individual with COVID-19 infection in the past 14 days at D-1.

   Physical and Laboratory Findings
10. Have a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus 1 and/or 2 antibodies (anti-HIV1 and anti HIV2 Ab) at screening.
11. Positive findings of urine drug screen (methadone, barbiturates, morphine, amphetamines, methamphetamines, opiates (including morphine), cannabinoids, cocaine, benzodiazepines, tricyclic antidepressants (TCA), 3,4-methylenedioxy-methamphetamine [MDMA; ecstasy]).
12. Have a positive alcohol breath test result at screening or D-1.

    Lifestyle restrictions
13. Have regular consumption of grapefruit juice and any xanthine-containing products (e.g., coffee, tea, chocolate, or Coca-Cola like drinks) more than 6 cups per day (or equivalent), or consumption of any alcoholic beverages within 48 h before prior dosing (D1) until final discharge day inclusive.
14. Have regular consumption of alcoholic beverages that exceeds 21 units per week (1 unit = 10 g of pure alcohol).

    Prior/Concurrent Clinical Study Experience
15. Participation in any another interventional study within ≤90 days prior to Screening provided that the clinical study did not entail administration of a biological compound with a long terminal phase half-life (t½), or in the exclusion period of a previous trial or participation in more than 3 clinical studies within the last 12 months.

    Prohibited Treatments
16. Use of any prescribed or non-prescribed drugs (including vitamins, herbal and dietary supplements, e.g., St. John's Wort) within 2 weeks or 5 half-lives, whichever is longer, prior to study drug administration, except for the occasional use of acetaminophen (up to 3 g/day).

    Other Exclusions
17. Subjects who, in the opinion of the Investigator, are not likely to complete the study for whatever reason.
18. Subject is employed by Sponsor, the CRO, or study site (permanent, temporary contract worker, or designee responsible for the conduct of the study) or is immediate family (i.e., a spouse, parent, sibling, or child, whether biological or legally adopted) of Sponsor, CRO, or study site employee.
19. Prisoners or subjects who are legally institutionalized and with right's restrictions.
20. For Part 1 SAD optional exploratory cohort with CSF sampling only:

    * Platelets and coagulation results within normal ranges.
    * Any medical history that could contraindicate a lumbar puncture [such as spinal trauma, scoliosis, regular headaches (non-exhaustive list)].
    * Use of aspirin or any anticoagulant medication within 3 weeks prior to CSF sampling

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Mâle
Enrollment: 92 (Actual)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single dose | From Day 1 to Day 7
  • Percentage of subjects who experienced at least one treatment-emergent adverse event (TEAE) by seriousness, intensity, and relatedness from baseline through follow-up,
Safety and tolerability of single dose | From Day 1 to Day 7
  • Percentage of subjects who discontinued due to a TEAE,
Safety and tolerability of single dose | From Day 1 to Day 7
  • Percentage of subjects who met the abnormal criteria for safety laboratory tests at least once post-dose,
Safety and tolerability of single dose | From Day 1 to Day 7
  • Percentage of subjects who met the abnormal criteria for vital signs (blood pressure, pulse rate, and body temperature) measurement at least once post-dose,
Safety and tolerability of single dose | From Day 1 to Day 7
  • Percentage of subjects who meet the abnormal criteria for safety electrocardiogram (ECG) parameters at least once post-dose.
Safety and tolerability of multiple dose | From Day 1 to Day 19
  • Percentage of subjects who experienced at least one treatment-emergent adverse event (TEAE) by seriousness, intensity, and relatedness from baseline through follow-up,
Safety and tolerability of multiple dose | From Day 1 to Day 19
  • Percentage of subjects who discontinued due to a TEAE,
Safety and tolerability of multiple dose | From Day 1 to Day 19
  • Percentage of subjects who met the abnormal criteria for safety laboratory tests at least once post-dose,
Safety and tolerability of multiple dose | From Day 1 to Day 19
  • Percentage of subjects who met the abnormal criteria for vital signs (blood pressure, pulse rate, and body temperature) measurement at least once post-dose,
Safety and tolerability of multiple dose | From Day 1 to Day 19
  • Percentage of subjects who meet the abnormal criteria for safety electrocardiogram (ECG) parameters at least once post-dose.

SECONDARY OUTCOMES:
SAD - Cmax | Day 1
  Maximum observed plasma concentration (Cmax)
SAD tmax | Day 1
  Time to reach maximum observed plasma concentration (tmax)
SAD Clast | Day 1
  Last observed quantifiable concentration (Clast)
SAD Tlast | Day 1
  Time to reach last observed quantifiable concentration (Tlast)
SAD AUC0-inf | Day 1
  Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf)
SAD AUC0-t | Day 1
  Area under the plasma concentration-time curve from time zero to time t (AUC0-t)
SAD ke | Day 1
  Apparent terminal elimination rate constant (ke)
SAD t½ | Day 1
  Terminal elimination half-life (t½)
SAD CL/F | Day 1
  Total body clearance (CL/F)
SAD Vz/F | Day 1
  Volume of distribution (Vz/F)
MAD Cmax | Day 1 and Day 12
  Maximum observed plasma concentration (Cmax)
MAD tmax | Day 1 and Day 12
  Time to reach maximum observed plasma concentration (tmax)
MAD Ctrough | Day 1 and Day 12
  Trough concentration at the end of the dosing interval (Ctrough)
MAD AUC0-24h | Day 1 and Day 12
  Area under the plasma concentration-time curve from time zero to 24h (AUC0-24h)
MAD AUC0-inf | Day 1 and Day 12
  Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf)
MAD ke | Day 1 and Day 12
  Terminal elimination constant rate (ke)
MAD t½ | Day 1 and Day 12
  Terminal elimination half-life (t½)
MAD CL/F | Day 1 and Day 12
  Total body clearance (CL/F)
Characterize MAD PK profiles of VNA-318 | Day 1 and Day 12
  Volume of distribution (Vz/F)
MAD Vss | Day 12
  Apparent volume of distribution at steady-state (Vss)
MAD accumulation ratio | Day 12
  Accumulation ratio calculated from Cmax at steady state and Cmax after first dosing (Rac(Cmax)) as well as from AUC (Rac(AUC(0-24h))

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Dugi, MD, Study Director — Vandria SA
Locations (1):
- Biotrial, Rennes, France

IPD SHARING:
Plan to Share IPD: No